CLINICAL TRIAL: NCT04808076
Title: Advanced MR-methods, Protein Levels in Cerebrospinal Fluid, Gait Analysis and Symptoms in Patients with Idiopathic Normal Pressure Hydrocephalus.
Brief Title: Idiopathic Normal Pressure Hydrocephalus: Focus on Imaging and Clinical Symptoms.
Acronym: LiNPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Fredrik Lundin, Senior Officer, MD, PhD, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LinkoepingU2
Record Dates: First submitted 2021-02-23; First posted 2021-03-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2023-03

CONDITIONS: Fecal Incontinence with Fecal Urgency; Urine Incontinence; Diffusion Tensor Imaging; Leukoencephalopathies
Keywords: Tract-Based Spatial Statistics; DTI; fecal incontinence; urine incontinence; whiter matter changes
MeSH Terms: conditions — Nocturnal Enuresis; Leukoencephalopathies; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: INPH patients and Healthy Individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iNPH patients (Active Comparator): Shunt operation
  Interventions: Procedure: Shunt surgery
- Healthy Individuals (No Intervention): Healthy individuals without any neurological disease.

INTERVENTIONS:
Procedure: Shunt surgery — Shunt operation
  Arms: iNPH patients

SUMMARY:
LiNPH is a prospective single center clinical and radiological study.

DETAILED DESCRIPTION:
Fifty consecutive patients with idiopathic Normal Pressure Hydrocephalus (iNPH) diagnosed according to the American-European iNPH guidelines from 2005, are going to be recruited from the outpatient clinic at the Department of Neurology, University Hospital, Linköping, Sweden. All patients are going to undergo a primary evaluation and examination by a neurologist followed by a CT or/and a MRI of the brain. On MRI there should be symmetrical communicating ventricular enlargement without cortical infarcts or other lesions of clinical importance, except lacunar infarcts (<1 cm3), the Evans ratio should be ≥ 0.3 and the corpus callosum angle should be between 50o to 90o. The temporal horns and third ventricle should be relatively enlarged. Mild to moderate cortical atrophy and subcortical white matter hyper-intensity will be allowed. The motor function will be assessed by a physiotherapist using the following tests: time needed for a 10-meter (m) walk in steps (w10ms) and 10-m walk in time (w10mt) at a self-selected speed and with their usual walking aid, timed up and go test in seconds (TUGt) and steps (TUGs), which is a timed test for standing up from chair, walking 3 m, turning and walking back to the chair and sitting down. An occupational therapist will perform cognitive testing with Mini Mental State Examination (MMSE). A CSF-tap-test will be performed at the Neurology outpatient department, at around 10:00 pm, in all patients. For the CSF-TT the patients will lie in a recumbent position, and under sterile conditions by using a 10 ml subcutaneous Xylocaine dose as pain prevention, the investigators will applicate a spinal needle 18Gx3.50"x1.2mmx90mm. Once CSF is obtained, a spinal fluid manometer (Optidynamic, Mediplast, Italy) will be connected to measure the CSF pressure in cm H2O. The lumbar pressure will be measured during a period of almost one minute for avoiding artificially elevated levels. All patients will be relaxed and have their neck to a neutral position and their legs extended. Lumbar pressure will be measured before the CSF-TT. The CSF will be analyzed for: cells, lactate, albumin, isoelectric focusing, antibodies against Borrelia Burgdofferi, NFL, t-tau, p-tau, β-amyloid 42/40, β-amyloid and GFAP. After a multidisciplinary round the investigators will decide who is suitable for a ventriculoperitoneal shunt. All probable/possible iNPH patients, included in the study, will undergo a preoperative Tracted-Based Spatial Statistics (TBSS) and Diffusion Tensor Imaging (DTI) investigation one to two days before the operation. All included in this study patients will undergo the same work-up almost 3 months after the shunt surgery inclusive the TBSS and DTI. All patients will meet a neurosurgeon once after the operation for possible shunt valve adjustment.

In addition, 50 volunteer healthy control subjects (HI) over the age of 60 will be recruited. All HI will undergo examination by a neurologist, DTI,TBSS and answer questionnaires included in the study. The controls are recruited from relatives, University Hospital employees and friends of the research group through advertising and personal inquiries. Exclusion criteria are observable gait disorder, diagnosed dementia, obvious gait / balance disorder for other reasons, occurrence of claustrophobia, implants that make MRI examination impossible and neurological disorder that is detected in connection with MRI examination and urinary catheter and / or uro- / intestinal stomia.

Another part of this project is a qualitative questionnaire based single center prospective study. All LiNPH patients and HI are going to answer three questionnaires ( ICIQ-UI, Bowel function Questionnaire, Wexners FI) regarding gastrointestinal and urinary symptoms and the investigators are going to correlate them with clinical data before and after the shunt surgery. The aim of this study is to identify if fecal incontinence is a new unknown symptom in iNPH patients. The secondary aim of this study is to correlate DTI and TBSS data with urinary- and fecal-incontinence symptoms.

The primary aim of this study is to distinguish between reversible and irreversible changes in iNPH. To establish a new technique in investigation of patients with iNPH and early identify this group. A significant correlation between DTI results in one or more brain areas with the iNPH-results will give the investigators the opportunity to use a specific DTI protocol to easier identify iNPH-patients who will have positive results with a shunt operation. The investigators also aim to compare manual-DTI MRI and TBSS-based MRI results before and after shunt surgery.

ELIGIBILITY:
Inclusion Criteria: Patients fulfilling the clinical and radiological criteria for a possible or probable iNPH diagnosis, according to the American-European Guidelines from 2005.

-

Exclusion Criteria: Patients unable to understand instructions with an MMSE lower than 17, claustrophobia or implant which makes the participation in MRI studies unable.

-

Ages: 61 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
White Matter Changes in Idiopathic Normal Pressure Hydrocephalus: A Diffusion Tensor Imaging Study. | 2 years
  Franctional Anisotropi and Apparent Diffusion Coefficient changes before and 3 months after the shunt surgery and correlation with clinical data. All data will be compared with results from the Healthy individual group.

SECONDARY OUTCOMES:
Gastrointestinal and urinary symptoms in idiopathic Normal Pressure Hydrocephalus. | 2 years
  By using questionnaires possible gastrointestinal and urinary symptoms are going to be characterized, check existence and correlate with Diffusion Tensor Imaging data. Statistically control of differences with the Healthy Individual group.

OTHER OUTCOMES:
Tract-based spatial statistics and diffusion tensor imaging in patients with idiopathic Normal Pressure Hydrocephalus. | 2 years
  Analysis of data from both techniques and statistical analysis to find which method could be more suitable in patients with idiopathic Normal Pressure Hydrocephalus.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Lundin, MD, PhD, Study Director — Department of Neurology and Department of Biomedical and Clinical Sciences, Linköping University
Locations (1):
- University Hospital of Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eleftheriou A, Blystad I, Tisell A, Gasslander J, Lundin F. Publisher Correction: Indication of Thalamo-Cortical Circuit Dysfunction in Idiopathic Normal Pressure Hydrocephalus: A Diffusion Tensor Imaging Study. Sci Rep. 2020 Jul 16;10(1):12014. doi: 10.1038/s41598-020-69149-x. PMID 32678296
- [Background] Keong NC, Pena A, Price SJ, Czosnyka M, Czosnyka Z, DeVito EE, Housden CR, Sahakian BJ, Pickard JD. Diffusion tensor imaging profiles reveal specific neural tract distortion in normal pressure hydrocephalus. PLoS One. 2017 Aug 17;12(8):e0181624. doi: 10.1371/journal.pone.0181624. eCollection 2017. PMID 28817574
- [Background] Siasios I, Kapsalaki EZ, Fountas KN, Fotiadou A, Dorsch A, Vakharia K, Pollina J, Dimopoulos V. The role of diffusion tensor imaging and fractional anisotropy in the evaluation of patients with idiopathic normal pressure hydrocephalus: a literature review. Neurosurg Focus. 2016 Sep;41(3):E12. doi: 10.3171/2016.6.FOCUS16192. PMID 27581308
- [Background] Nakanishi A, Fukunaga I, Hori M, Masutani Y, Takaaki H, Miyajima M, Aoki S. Microstructural changes of the corticospinal tract in idiopathic normal pressure hydrocephalus: a comparison of diffusion tensor and diffusional kurtosis imaging. Neuroradiology. 2013 Aug;55(8):971-976. doi: 10.1007/s00234-013-1201-6. Epub 2013 Jun 2. PMID 23728069
- [Background] Ege S. [Management of urinary incontinence in a geriatric rehabilitation department : Global urinary incontinence assessment incorporating the International Consultation on Incontinence Questionnare - Urinary Incontinence Short Form (ICIQ-UI SF)]. Z Gerontol Geriatr. 2018 Apr;51(3):301-313. doi: 10.1007/s00391-016-1173-3. Epub 2017 Feb 8. German. PMID 28180932
- [Background] Marmarou A, Black P, Bergsneider M, Klinge P, Relkin N; International NPH Consultant Group. Guidelines for management of idiopathic normal pressure hydrocephalus: progress to date. Acta Neurochir Suppl. 2005;95:237-40. doi: 10.1007/3-211-32318-x_48. PMID 16463856
- [Background] Ishikawa M, Hashimoto M, Kuwana N, Mori E, Miyake H, Wachi A, Takeuchi T, Kazui H, Koyama H. Guidelines for management of idiopathic normal pressure hydrocephalus. Neurol Med Chir (Tokyo). 2008;48 Suppl:S1-23. doi: 10.2176/nmc.48.s1. PMID 18408356